CLINICAL TRIAL: NCT04754087
Title: Global, Multicenter, and Prospective Post-Market Clinical Follow-Up Study of the G7 Acetabular System With Vivacit-E and Longevity Highly Crosslinked Polyethylene (HXLPE) Liners & Instrumentation
Brief Title: G7 Acetabular System With Vivacit-E or Longevity Liner PMCF Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMG2019-32H
Record Dates: First submitted 2021-01-25; First posted 2021-02-15 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Total Hip Arthroplasty; Degenerative Joint Disease of Hip; Avascular Necrosis of Hip; Rheumatoid Arthritis of Hip; Osteoarthritis, Hip; Osteoarthritis of Hip; Fractures, Hip; Fracture of Hip
MeSH Terms: conditions — Osteoarthritis, Hip; Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- G7 Shell with Vivacit-E and Longevity Highly Crosslinked Polyethylene Liners (Other): Up to 300 hips globally will be implanted with a G7 Shell and either the Vivacit-E or Longevity Liner. The liner used by each site will be identified at start-up.
  Interventions: Device: Vivacit-E and Longevity (HXLPE) Liners

INTERVENTIONS:
Device: Vivacit-E and Longevity (HXLPE) Liners — This is a dual cohort study in which 150 subjects will receive the Vivacit-E (HXLPE) Liner and 150 subjects will receive the Longevity (HXLPE) Liner.

SUMMARY:
The main objectives of this study are to confirm the long-term safety, performance, and clinical benefits of the G7 Acetabular Shells when used with the Vivacit-E and Longevity HXLPE liners and instrumentation in primary and revision total hip arthroplasty.

DETAILED DESCRIPTION:
The primary endpoint is defined by the survival of the implant system at 10 years, which is based on removal or intended removal of the study device and will be determined using Kaplan Meier method. The safety of the system will be assessed by monitoring the frequency and incidence of adverse events. Relation of the events to either implant or instrumentation should be specified.

The secondary endpoints are the assessment of performance and clinical benefits by recording patient-reported clinical outcomes measures (PROMs) as well as radiographic outcomes (if available).

ELIGIBILITY:
Inclusion Criteria:

* Patient must be a legal adult who has reached full skeletal maturity.
* Patient must be treated for one of the following indications:
* Noninflammatory degenerative joint disease including osteoarthritis and avascular necrosis
* Rheumatoid arthritis
* Correction of functional deformity
* Treatment of non-union, femoral neck fracture, and trochanteric fractures of the proximal femur with head involvement, unmanageable by other techniques
* Revision procedures where other treatment or devices have failed
* Patient must be able and willing to complete the protocol required follow-up visits.
* Patient must be able and willing to sign the Institutional Review Board or Ethics Committee (IRB/EC) approved informed consent.

Exclusion Criteria:

* Patient presents with osteoporosis, which in the opinion of the Principal Investigator, may limit the subject's ability to support total hip arthroplasty using the study device.
* Patient has a metabolic disorder that may impair bone formation.
* Patient has osteomalacia.
* Patient has distant foci of infections which may spread to the implant site or patient with infection, sepsis or osteomyelitis.
* Patient has rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram.
* Patient has a vascular insufficiency, muscular atrophy, or neuromuscular disease
* Patient is a prisoner.
* Patient is a current alcohol or drug abuser.
* Uncooperative patient or patient with neurologic disorders who is incapable or unwilling to follow directions.
* Patient is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival of the study device (liner); whether or not it is still implanted in the subject | At 10 years
  Survivorship will be based on revision or intended revision of the study device (liner).
Adverse Event (safety) | At 10 years
  Safety will be evaluated by monitoring the frequency and incidence of device related adverse events or unanticipated adverse device effects in investigational subjects.

SECONDARY OUTCOMES:
Pain and Function using Modified Harris Hip Score | At 10 years
  Pain and function will be measured using the Modified Harris Hip Score self assessment. The overall score runs from 0-100 with 100 representing the best outcome.
Pain and Function using Oxford Hip Score | At 10 years
  Pain and function will be measured using the Oxford Hip Score self assessment. The overall score runs from 0-48 with 48 representing the best outcome.
Patient Quality of Life using EQ-5D-5L Descriptive System | At 10 years
  Perceived qualify of life will be measured using the EQ-5D-5L Descriptive System - comprises mobility, self care, usual activities, pain/discomfort, anxiety/depression. Each question in this section has an overall score of 1-5 with 1 representing the best health.
Patient Quality of Life using EQ-5D-5L EQ visual analogue scale | At 10 years
  Perceived qualify of life will be measured using the EQ visual analogue scale (EQ VAS) - records the respondent's self-rated health on a vertical, visual analogue scale. This section has an overall score of 0-100 with 100 representing the best health.

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, Study Director — Zimmer Biomet
Locations (11):
- United States (6):
  - Colorado Joint Replacement, Denver, Colorado
  - South Bend Orthopaedics, South Bend, Indiana
  - Duke University Medical Center, Durham, North Carolina
  - Slocum Center for Orthopedics & Sports Medicine, Eugene, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - University of Utah Health, Salt Lake City, Utah
- Copenhagen University Hospital Hvidovre, Hvidovre, Denmark
- Netherlands (2):
  - Zuyderland Hospital, Geleen
  - OCON Hengelo, Hengelo
- Skane University Hospital, Lund, Sweden
- The Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust Royal Bournemouth Hospital, Bournemouth, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No